CLINICAL TRIAL: NCT01205308
Title: Effects of Plant Stanol Esters on Serum Lipids, Precursors of Cholesterol Synthesis and Plant Sterols in Type 1 Diabetics on Stabile Statin Drug Use
Brief Title: Plant Stanols and Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: Kuopio University Hospital (Other); Raisio Plc (Industry)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 125/2009
Record Dates: First submitted 2010-09-13; First posted 2010-09-20 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Type 1 Diabetes
Keywords: Plant stanols; type 1 diabetes; sterol metabolism; cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stanol ester spread (Active Comparator): Vegetable oil based margarine with stanol ester enrichment
  Interventions: Dietary Supplement: Vegetable oil based margarine with plant stanol ester enrichment
- control spread (Placebo Comparator): Vegetable oil based margarine without stanol ester enrichment
  Interventions: Dietary Supplement: Vegetable oil based margarine with plant stanol ester enrichment

INTERVENTIONS:
Dietary Supplement: Vegetable oil based margarine with plant stanol ester enrichment — 3 g plant stanols/ day

SUMMARY:
In type 1 diabetes (T1D) coronary artery disease (CAD) is an important cause of morbidity and mortality. Although serum cholesterol concentrations are not always elevated in T1D, cholesterol metabolism is different from non-diabetics, so that cholesterol absorption is enhanced. The aim of this study is to investigate the effects of plant stanol esters on serum lipid and lipoprotein lipid concentrations, plant sterol and cholestanol concentrations as well as cholesterol metabolism in T1 diabetics on statin use. The study will give new information about how addition of plant stanol esters on statin use improve hypolipidemic effects in type 1 diabetes.

DETAILED DESCRIPTION:
In type 1 diabetes (T1D) coronary artery disease (CAD) is an important cause of morbidity and mortality. Although serum cholesterol concentrations are not always elevated in T1D, cholesterol metabolism is different from non-diabetics, so that cholesterol absorption is enhanced. Thus, theoretically, the best way to reduce serum cholesterol concentrations is to reduce cholesterol absorption. However, statins are recommended to T1 diabetics at the same LDL cholesterol levels as for type 2 diabetics to reduce risk to CAD.

The aim of this study is to investigate the effects of plant stanol esters on serum lipid and lipoprotein lipid concentrations, plant sterol and cholestanol concentrations as well as cholesterol metabolism in T1 diabetics on statin use.

Altogether, twenty-four T1 diabetics (HbA1c <9%) on stabile statin use will be recruited to the study from an announcement in the local newspaper and from Kuopio University Hospital and Harjula Hospital. The study is carried out with a randomized, double-blind and parallel design. The intervention group (n=12) consumes spread enriched with plant stanol esters (3 g/d stanols) and the control group (n=12) the same spread containing no added stanols for 4 weeks. The fasting blood samples are taken at weeks 0, 3 and 4. From blood samples concentrations of serum lipids, squalene and non-cholesterol sterols will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes, stabile statin drug use, HbA1c <9%

Exclusion Criteria:

* liver, kidney and thyroid dysfunction, severe diabetic proteinuria, gastroparesis, unstable CAD, unstable inflammatory gastrointestinal disease

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
serum lipids | Week 0
serum lipids | Week 3
serum lipids | Week 4
squalene | Week 0
squalene | Week 3
squalene | Week 4
non-cholesterol sterols | Week 0
non-cholesterol sterols | Week 3
non-cholesterol sterols | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gylling, Professor, Study Director — University of Eastern Finland; Maarit Hallikainen, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland